CLINICAL TRIAL: NCT04962932
Title: Internet-delivered Cognitive Behavior Therapy Compared to Stress Management for Atrial Fibrillation- a Randomized Controlled Trial With Active Control
Brief Title: Internet-delivered Cognitive Behavior Therapy Compared to Stress Management for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate professor,PhD, Lic. psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF RCT 2
Record Dates: First submitted 2021-06-24; First posted 2021-07-15 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Arrythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered exposure-focused CBT (Experimental): Internet-delivered CBT over 10 weeks The CBT treatment lasts for 10 weeks and includes the following: Education on the role of anxiety on cardiac function and the effects of symptom preoccupation and avoidance QoL and depression in AF, creating a vicious cycle; exposure to physical sensations that are similar to AF symptoms (e.g.,palpitations due to physical activity or stress) to reduce fear of these symptoms; exposure to situations or activities previously avoided and abolishment of behaviors that aim to control symptoms; and behavioral activation aiming to increase social and physical activity and reduce depressive symptoms. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internet-deliviered exposure-based CBT
- Internet-delivered stress management treatment (Active Comparator): Stress management treatment for 10 weeks Participants randomized to The Stress Management Treatment will receive 10 weeks of stress managemen including relaxation technics, standard life style advice regarding physical activity, sleep and and standardized AF-information in line with current guidelines for AF. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internet-delivered stress management treatment

INTERVENTIONS:
Behavioral: Internet-deliviered exposure-based CBT — The intervention lasts for 10 weeks and include: Education, Interoceptive exposure, exposure in-vivo, combining in-vivo exposure with interoceptive exposure, behavioral activation and relapse prevention. Include the guidance of a minimum weekly contact with a CBT psychologist.
  Arms: Internet-delivered exposure-focused CBT
Behavioral: Internet-delivered stress management treatment — The intervention last for 10 weeks and include: Internet-SMT include life-style advice (e.g., exercise, sleep advice), relaxation and problem-solving skills to reduce stress. Patients are offered regular online contact with a psychologist with the same frequency and intensity as in the CBT arm.
  Arms: Internet-delivered stress management treatment

SUMMARY:
The aim of this study is to evaluate if internet- delivered cognitive behavior therapy (CBT), based on exposure principles and behavioral activation, improves QoL and symptom burden in patients with symptomatic atrial fibrillation (AF), controlling for expectancy of improvement and attention from a caregiver, using an active control group (stress management). The study will include 260 patients with symptomatic AF despite optimal medical treatment in accordance with current guidelines.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia (irregular heartbeat) affecting 3% of the population. AF is associated with poor quality of life (QoL) and large costs for society. In a considerable proportion of patients, AF symptoms (e.g., palpitations, fatigue, and chest pain) are not alleviated by current medical or interventional treatments. Psychological factors can worsen AF symptoms, and anxiety and depression are common among AF patients. Symptom preoccupation and avoidance of social and physical activities are likely to play important roles in the development of anxiety, depression, disability and healthcare utilization.

The aim is to evaluate if CBT, based on behavioral activation and exposure principles, improves wellbeing and QoL in symptomatic AF patients controlling for expectancy of improvement and attention from a caregiver using an active control group receiving stress management treatment (SMT).

Method: A randomized controlled trial. Participants are randomized to internet- delivered exposure-based CBT (N=130) or to SMT (N=130). Participants in both groups receive weekly therapist support through online written communication. The internet-delivered SMT-treatment includes life-style advice (e.g., exercise, sleep advice), relaxation and problem-solving skills to reduce stress. Both treatments lasts 10 weeks and are comparable regarding number of treatment modules, treatment burden and attention from the treating psychologist.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal AF ≥ once per month that causes moderate to severe symptoms and leads to significant distress or interferes with daily life (i.e. EHRA class ≥ IIb);
* Scoring ≥ 20 on the Cardiac Anxiety Questionnaire at screening;
* Age 18-75 years;
* On optimal medical treatment;
* Able to read and write in Swedish.

Exclusion Criteria:

* Heart failure with severe systolic dysfunction (ejection fraction ≤ 35%);
* Significant valvular disease;
* Planned ablation for AF or ablation within 3 months before assessment;
* Other severe medical illness;
* Any medical restriction to physical exercise;
* Severe psychiatric disorder, severe depression, or risk of suicide;
* Alcohol dependency;
* Previous participation in any AF-CBT study conducted by the research group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Effect on Quality-of-Life modified for weekly assessment | Change over 11 measurement points measured from baseline and weekly for 10 weeks during treatment [PRIMARY ENDPOINT]
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction. Total score ranges from 0 (severe symptoms and disability) to 100 (no symptoms and disability).
Atrial Fibrillation Effect on Quality-of-Life modified for weekly assessment | From baseline to 9 months
  The AFEQT is an atrial fibrillation-specific measure that taps into the QoL-domains: symptoms, daily activities, treatment concern, and treatment satisfaction. Total score ranges from 0 (severe symptoms and disability) to 100 (no symptoms and disability).

SECONDARY OUTCOMES:
Cardiac Anxiety Questionnaire (CAQ) | From baseline to 10 weeks
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac Anxiety Questionnaire (CAQ) | From baseline to 9 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
AF-avoidance behavior questionnaire | From baseline to 10 weeks
  Form measuring AF-specific avoidance- and control behaviors, developed by the research group
AF-avoidance behavior questionnaire | From baseline to 9 months
  Form measuring AF-specific avoidance- and control behaviors, developed by the research group
AF-avoidance behavior questionnaire modified for weekly assessment | Change over 11 measurement points measured from baseline and weekly for 10 weeks during treatment
  4 items from the AF-avoidance behavior questionnaire
Short Form Health Survey (SF-12) | From baseline to 10 weeks
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Short Form Health Survey (SF-12) | From baseline to 9 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Atrial Fibrillation Severity Scale (4 items) | From baseline to 10 weeks
  4 items from the Atrial Fibrillation Severity Scale, measuring health care seeking
Atrial Fibrillation Severity Scale (4 items) | From baseline to 9 months
  4 items from the Atrial Fibrillation Severity Scale, measuring health care seeking
The Godin-Shepard Leisure-Time Physical Activity Questionnaire | From baseline to 10 weeks
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
The Godin-Shepard Leisure-Time Physical Activity Questionnaire | From baseline to 9 months
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
Body Sensation Questionnaire | From baseline to 10 weeks
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | From baseline to 9 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Patient Health Questionnaire-2 | From baseline to 10 weeks
  Short form measuring depression, score ranging 0 to 6 with a higher score indicating higher level of depression.
Patient Health Questionnaire-2 | From baseline to 9 months
  Short form measuring depression, score ranging 0 to 6 ,with a higher score indicating higher level of depression.
Perceived Stress Scale (4 items version) | From baseline to 10 weeks
  Measures perceived stress, score ranging from 0-16, with a higher score indicating higher level of perceived stress
Perceived Stress Scale (4 items version) | From baseline to 9 months
  Measures perceived stress, score ranging from 0-16, with a higher score indicating higher level of perceived stress
Generalized Anxiety Disorder-2 (GAD-2) | From baseline to 10 weeks
  General anxiety, score ranging from 0-6, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder-2 | From baseline to 9 months
  General anxiety, score ranging from 0-6, with a higher score indicating more anxiety and worry.
Insomnia Severity Index (5 items) | From baseline to 10 weeks
  Measure of insomnia, score ranging from 0-20, with a higher score indicating more severe insomnia
Insomnia Severity Index (5 items) | From Baseline to 9 months
  Measure of insomnia, score ranging from 0-20, with a higher score indicating more severe insomnia
Perceived Competence Scale | From baseline to 10 weeks
  Perception of AF-specific knowledge and competence, score ranging from 0- 50 with higher score indicating higher perceived competence
Perceived Competence Scale | From baseline to 9 months
  Perception of AF-specific knowledge and competence, score ranging from 0- 50 with higher score indicating higher perceived competence
Client Satisfaction Questionnaire | 10 weeks from baseline
  Treatment satisfaction, score ranging from 0-24, with a higher score indicating higher satisfaction with treatment.
Adverse events | 10 weeks from baseline
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | 9 months from baseline
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Symptoms Checklist Severity and Frequency Scale (SCL) | From baseline to 10 weeks
  AF-related symptoms
Symptoms Checklist Severity and Frequency Scale (SCL) | From baseline to 9 months
  AF-related symptoms measured in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
AFFS/SCL-4 | Weekly from baseline to 10 weeks
  4 items derived from the Symptoms Checklist (SCL) and the Atrial Fibrillation Severity Scale (AFSS) measuring disabling cardiac symptoms not specified in AFEQT
AFFS/SCL-4 | From baseline to 9 months
  4 items derived from the Symptoms Checklist (SCL) and the Atrial Fibrillation Severity Scale (AFSS) measuring disabling cardiac symptoms not specified in AFEQT

OTHER OUTCOMES:
Psychosocial stressors and changes in physical health | 10 weeks from baseline
  Participants are asked about their self-perceived health and if they have experienced any stressful event that they believe have affected their health (e.g severe disease, death of close relative, divorce)
Psychosocial stressors and changes in physical health | 9 months from baseline
  Participants are asked about their self-perceived health and if they have experienced any stressful event that they believe have affected their health (e.g severe disease, death of close relative, divorce)
Background data | Baseline
  Demographics, list of medications, co-morbidity, smoking history and alcohol consumption
Treatment Credibility Scale | 2-4 weeks from baseline
  Measures treatment credibility
Working Alliance Inventory | 2-4 weeks from baseline
  Measures therapeutic alliance with the psychologist
Changes in medication | 10 weeks from baseline
  Participants are asked if they have made any changes in medication
Changes in medication | 9 months from baseline
  Participants are asked if they have made any changes in medication

CONTACTS AND LOCATIONS:
Overall Officials: Brjann Ljotsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska universitetssjukhuset Solna, Solna, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04962932/SAP_000.pdf